CLINICAL TRIAL: NCT02993315
Title: A Randomized, Double--blind, Placebo-controlled Phase III Study to Evaluate Active Immunization in Adjuvant Therapy of Patients with Stage IIIB and IIIC Melanoma with Natural Dendritic Cells Pulsed with Synthetic Peptides.
Brief Title: Melanoma Patients Immunized with Natural DenDritic Cells
Acronym: MIND-DC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch National Health Care Institute (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL55823.000.15
Record Dates: First submitted 2016-11-23; First posted 2016-12-15 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2022-04

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- nDC vaccination arm (Experimental): Patients in the nDC vaccination arm will receive a maximum of 3 cycles each consisting of 3 nDC injections intranodally (3-8x10^6 nDC).
  Interventions: Biological: nDC vaccination
- placebo arm (Placebo Comparator): Patients will receive a maximum of 3 cycles each consisting of 3 placebo injections intranodally.
  Interventions: Biological: placebo injection

INTERVENTIONS:
Biological: nDC vaccination
  Arms: nDC vaccination arm
Biological: placebo injection
  Arms: placebo arm

SUMMARY:
The aim of this study is to determine whether adjuvant treatment with nDC vaccination, after complete radical lymph node dissection or sentinel node procedure in stage IIIB and IIIC melanoma patients, improves recurrence-free survival (RFS) as compared to treatment with matching placebo.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, interventional study of nDC vaccination versus placebo. Dendritic cell-based immunotherapy consists of antigen-loaded autologous DC that are administered to patients with the intention of inducing antigen-specific T and B cell responses and proved safe with minimal side effects. Natural DC (nDC) consist of plasmacytoid DC and myeloid DC. Subjects will be randomized 2:1 and stratified by stage of disease, adjuvant radiotherapy, BRAF mutation status, HLA-type and nDC production centre. The treatment will be continued for a maximum of 1.5 years or until recurrence of disease, unacceptable toxicity or withdrawal from the study.

ELIGIBILITY:
Eligibility Criteria:

* at least 18 years of age.
* Histologically confirmed stage III cutaneous melanoma, classified as IIIB or IIIC disease (AJCC 2009). Patients with completely resected in-transit and/or satellite metastases and patients with unknown primary melanoma are allowed in this trial.
* Radical lymph node dissection involved site with complete resection or sentinel node procedure (in case of patients without RLND because of limited sentinel-node positive disease) of melanoma as documented on the operating report and pathology report with at least the minimal levels excised as stated in national guidelines.
* Radical lymph node dissection involved site with complete resection or sentinel node procedure (in case of patients without RLND because of limited sentinel-node positive disease) must be performed within 12 weeks prior to start of study.
* Recovered from definitive surgery (e.g. no uncontrolled wound infections or indwelling drains).
* Absence of distant metastases must be documented by a CT scan of the chest and abdomen (including pelvis) or a Positron Emission Tomography (PET) scan, the scan should have been performed within 6 weeks before surgery or after surgery prior to inclusion. In addition, a physical exam after surgery must be performed also excluding distant metastases.
* No clinical evidence for brain metastasis. If brain metastases are clinically suspected, a CT or Magnetic Resonance Imaging (MRI) scan of the brain must exclude brain metastases.
* World Health Organization (WHO) performance status of 0 or 1 at time of randomization.
* Adequate hematologic, renal and liver function as defined by laboratory values performed within 4 weeks of randomization.
* No second malignancy in the previous 5 years, with the exception of adequately treated carcinoma in-situ and basal or squamous cell carcinoma of the skin.
* No concomitant use of immunosuppressive drugs orally or intravenously. Topical and intranasal steroids are permitted.
* No uncontrolled infectious disease, i.e. negative testing for HIV, HBV, HCV and syphilis.
* No autoimmune disease such as, but not limited to, inflammatory bowel disease, multiple sclerosis, and lupus. Patients with type 1 diabetes mellitus, hypothyroidism after autoimmune thyroiditis and skin disorders are not excluded.
* No serious (bleeding and clotting) condition that may interfere with safe leukapheresis.
* No pregnant or lactating women.
* No Women Of Child-Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for up to 8 weeks after the last administration of the treatment. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea > 12 consecutive months].
* Patients must have absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions must be discussed with the patient before registration in the trial.
* Expected adequacy of follow-up.
* Written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2024-01 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival rate | 2 years
  The primary objective of this study is to determine whether adjuvant nDC vaccination, after complete radical lymph node dissection or sentinel node procedure in stage IIIB and IIIC melanoma patients, improves 2-year RFS rate as compared to treatment with matching placebo. Defined as the percentage of patients who are alive and without recurrence of melanoma 2 years after randomization.
Treatment of melanoma patients | The primary endpoint, 2-year RFS. At data cutoff, the median duration of follow-up was 56.3 months.
  Adjuvant treatment with nDC vaccination or placebo, after standard treatment

SECONDARY OUTCOMES:
Overall survival | 2-years and median
  Overall survival
Tumor specific T-cell response | week 1, week 9, week 10, week 31, week 39, week 57, week 65, week 78, month 24, month 60
  Tumor specific T-cell response
Quality of Life Questionnaires | baseline, week 14, week 26, month 12, month 24, month 36, month 60
  Quality of Life Questionnaires
Costs (direct and indirect) of treatment | 2 years
  Costs (direct and indirect) of treatment
QALY | 2 years
  A cost-effectiveness acceptability curve will be derived that is able to evaluate efficiency by using different tresholds (willingness to pay) for a QALY.
Adverse Events related to treatment | 1,5 year
  Adverse Events related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jolanda de Vries, Prof. dr., Principal Investigator — Radboud University Medical Center
Locations (5):
- Netherlands (5):
  - NKI-AvL, Amsterdam
  - VUmc, Amsterdam
  - Radboudumc, Nijmegen
  - ErasmusMC, Rotterdam
  - Isala klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided